CLINICAL TRIAL: NCT04413955
Title: Seraph®-100 Microbind® Affinity Blood Filter for the Treatment of COVID-19 Under Emergency Use Authorization: Data Registry
Brief Title: Registry of Seraph®-100 Microbind® Affinity Blood Filter for COVID-19 Under EUA
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: ExThera Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 001-Seraph®-100 for SARS-CoV-2
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Seraph®-100 Microbind® Affinity Blood Filter — Use of an extracorporeal broad-spectrum sorbent hemoperfusion filter to removed SARS-CoV-2 virus and circulating cytokines from the blood
  Other Names: Seraph

SUMMARY:
Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) has caused a global pandemic and is associated with significant morbidity and mortality. The mortality rate for COVID-19 patients admitted to an intensive care unit (ICU) who require mechanical intubation is approximately 75%. While the pathophysiology of severe COVID-19 has yet to be fully understood, it is possible that a combination of high viral loads and an overactive dysregulated inflammatory response may contribute. Therefore, the clearance of SARS-CoV-2 virus and cytokines could provide a more opportunistic environment for the innate immune system to clear the virus and establish lasting immunity. The Seraph®-100 Microbind® Affinity Blood Filter (Seraph®-100) is an extracorporeal broad-spectrum sorbent hemoperfusion filter for removing virus and cytokines from the blood. The FDA authorized an Emergency Use Authorization (EUA) for treatment of severe COVID-19 with the Seraph®-100. As part of the EUA, this registry study will collect de-identified data to assess safety and efficacy on the use of Seraph®-100 Microbind® Affinity Blood Filter in the treatment of COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 infection
* Confirmed or imminent respiratory failure
* At least one of the following conditions

  1. Early acute lung injury (ALI) or early acute respiratory distress syndrome (ARDS)
  2. Severe disease, defined as:

     * dyspnea,
     * respiratory frequency ≥ 30 bpm,
     * blood oxygen saturation ≤ 93%,
     * partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, and/or
     * lung infiltrates > 50% within 24 to 48 hours
  3. Life-threatening disease, defined as:

     * respiratory failure,
     * septic shock, and/or
     * multiple organ dysfunction or failure

Exclusion Criteria:

* No Exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients in intensive care units in the US
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of known, expected, or unanticipated adverse device effects | From the initiation of therapy through 24 hours after therapy has been completed
  Monitor and report on adverse events and unanticipated adverse device effects experienced by patients receiving treatment with the Seraph®-100 for COVID-19, including but not limited to: bleeding, clotting, cardiac dysrhythmia, hypotension, increase in oxygen requirement, hemolytic anemia, and allergic/anaphylactic reaction

SECONDARY OUTCOMES:
Change in cardiovascular hemodynamic stability | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in Mean Arterial Pressure before and after treatment with the Seraph®-100 device
Change in cardiovascular hemodynamic support | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in required Vasopressor Dosages before and after treatment with the Seraph®-100 device
Change in pulmonary/respiratory status | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in required Respiratory Support before and after treatment with the Seraph®-100 device
Change in laboratory measures of cytokine reactions and/or viral sepsis: IL-6 | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in Interleukin-6 (IL-6) before and after treatment with the Seraph®-100 device
Change in laboratory measures of cytokine reactions and/or viral sepsis: CRP | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in C-Reactive Protein (CRP) before and after treatment with the Seraph®-100 device
Change in laboratory measures of cytokine reactions and/or viral sepsis: Ferritin | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in Ferritin before and after treatment with the Seraph®-100 device
Change in laboratory measures of cytokine reactions and/or viral sepsis: D-Dimer | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in D-Dimer before and after treatment with the Seraph®-100 device
Change in laboratory measures of cytokine reactions and/or viral sepsis: ALC | 24 hours prior to therapy through 24 hours after therapy has been completed
  Measure change in Absolute Lymphocyte Count (ALC) before and after treatment with the Seraph®-100 device

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Sun X, Yang S, Al-Dossary AA, Broitman S, Ni Y, Guan M, Yang M, Li J. Nanobody-Functionalized Cellulose for Capturing SARS-CoV-2. Appl Environ Microbiol. 2022 Mar 8;88(5):e0230321. doi: 10.1128/aem.02303-21. Epub 2022 Jan 5. PMID 34985974